CLINICAL TRIAL: NCT06084000
Title: STrategies of Scheduled Drug-coated Balloons (DCB) Versus Conventional DES for the interveNTional Therapy of de Novo Lesions in Large Coronary vESSels (STENTLESS) Trial
Acronym: STENTLESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Yongjian Wu, MD, PhD, Director of Coronary Heart Disease Center, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-I2M-1-002
Record Dates: First submitted 2023-09-26; First posted 2023-10-16 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Drug-coated Balloon; Drug-eluting Stent; De Novo Stenosis
MeSH Terms: interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-coated balloon dominant strategy (Experimental): * Patients will receive DCB (Bingo©, Yinyi Ltd., China) only if pre-dilation of the lesion was successful, or otherwise receive bailout stenting.
  * If bailout stenting is indicated, patients will receive any type of commercially available 2nd Gen DES at physician's preference.
  Interventions: Device: Drug-coated balloon (Bingo© [Paclitaxel-coated Balloon], Yinyi Ltd., China)
- Drug-eluting stent only strategy (Active Comparator): -For conventional stenting, patients will receive any type of commercially available 2nd Gen DES at physician's preference.
  Interventions: Device: Drug-eluting stent

INTERVENTIONS:
Device: Drug-coated balloon (Bingo© [Paclitaxel-coated Balloon], Yinyi Ltd., China) — * Patients treated with DCB will receive dual antiplatelet therapy (DAPT, aspirin plus P2Y12 inhibitor) for 1-3 months, followed by long-term single antiplatelet therapy (SAPT, aspirin or P2Y12 inhibitor).
  * Patients with bailout stenting will generally receive DAPT for 6 months unless deemed as with high ischemic and/or bleeding risks (see "special consideration" in Drug-eluting stent Arm), and then followed by long-term SAPT.
  Arms: Drug-coated balloon dominant strategy
Device: Drug-eluting stent — * Patients treated with DES will generally receive DAPT for 6 months unless deemed as with high ischemic and/or bleeding risks (see "special consideration" below), and then followed by long-term SAPT.
  * Special consideration:
    1. Patients will take additional assessment (both DAPT score and PRECISE-DAPT score) to determine their personalized duration of DAPT.
    2. The duration of DAPT is extended to 12 months for patients diagnosed as acute coronary syndrome within 12 months.
    3. If anticoagulation is indicated, patient will receive a short-term triple antithrombotic therapy (generally 1 to 4 weeks), followed by a variable length of dual antithrombotic therapy (oral anticoagulation (OAC) plus a single antiplatelet agent, preferably clopidogrel) and subsequent long-term OAC mono-therapy. The duration of dual antithrombotic therapy is determined by bleeding risks (HAS-BLED score) according to current guidelines.
  Arms: Drug-eluting stent only strategy

SUMMARY:
This is a multicenter, open-label, randomized controlled study meant to compare the safety and efficacy of scheduled drug-coated balloon (DCB) and conventional drug-eluting stent (DES) strategy in the treatment of de novo lesions of large coronary vessel with diameter larger than 2.75 mm. The trial was designed to provide high-quality evidence for expanding the clinical indications of DCB, and to explore a better way for coronary intervention based on DCB.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* De novo lesions of large coronary vessels with the diameter of target lesion reference vessel > 2.75 mm
* Single- or multi-vessel disease with only 1 lesion meeting the definition of severe stenosis and anatomically amenable to coronary revascularization using DCB alone judged by physician.

  * Severe stenosis is defined if 1 of the following criteria are met:

    1. visual angiographic stenosis with severity >= 70%.
    2. functional stenosis with quantitative flow reserve (QFR) or fractional flow reserve (FFR) < 0.8.
* Other coronary artery lesions are not recommended for coronary revascularization by current guidelines and are not likely need to be treated within the next 1 year judged by physician (e.g., visual stenosis with severity between 50-70% and FFR > 0.8)
* The prospective subject is agreed on participating the study with a formal written consent

Exclusion Criteria:

* History of acute coronary syndrome within the last 6 months.

  * Acute coronary syndrome is defined as 1 of following diagnosis:

    1. Unstable Angina Pectoris (UAP)
    2. ST-Elevated Myocardial Infarction (STEMI)
    3. Non-ST-Elevated Myocardial Infarction (NSTEMI)
  * Diagnosis of myocardial infarction (MI) requires both clinical evidence of myocardial ischemia and elevation of cardiac Troponin (cTn) I or T values with at least 1 value above the 99th percentile upper normal range limit (URL)
  * Clinical evidence of myocardial ischemia is defined as 1 of the following:

    1. Symptoms of myocardial ischemia
    2. New ischemic ECG changes
    3. Development of pathological Q waves
    4. Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischemic etiology
    5. Identification of a coronary thrombus by angiography
  * All types of MI (type 1 to 5 MI) defined by "the Fourth Universal Definition of Myocardial Infarction (2018)", which occurred within the last 6 months from inclusion phase would be excluded from this study.
* Patients who have received percutaneous coronary intervention (including stent implantation, plain old balloon angioplasty, and DCB angioplasty) within 12 months before the index procedure.
* Currently recommended indications for DCB: in-stent restenosis, bifurcation lesions requiring concomitant intervention of the major vessel and its adjacent side branch (e.g., lesions requiring dual stent implantation, kissing balloon technique, etc.)
* Lesions with any of the following anatomical characteristics presumably not suitable for DCB treatment:

  1. long lesion with length >= 40mm.
  2. severely calcified, moderate or severe tortuous, or severe angulated vessels, especially when vessel recoil seems possible.

     * Moderate tortuosity: 2 bends >75° or 1 bend >90° to reach the target lesion.
     * Severe tortuosity: 2 bends >90° or 3 bends >75° to reach the target lesion.
     * Severe angulation: angulated segment > 90°
     * Severe calcification: radiopacities noted without cardiac motion before contrast injection generally compromising both sides of the arterial lumen
  3. Chronic total occlusion

     * Definition: A lesion of a coronary artery becomes completely blocked for a duration of greater than or equal to 3 months based on angiographic evidence.
  4. lesions in left main coronary artery
  5. lesions in venous or arterial graft
* Chronic heart failure with left ventricular ejection fraction < 35% after 6 months of Guideline-Directed Medical Treatment (GDMT)
* Acute heart failure, hemodynamic instability, or cardiogenic shock

  * Acute heart failure is defined as a rapid onset of new or worsening signs and symptoms of heart failure.
* Non-cardiac Comorbidities:

  1. Severe liver insufficiency defined as 1 of the following:

     * alanine transaminase or aspartate transaminase more than 5-fold of upper reference limit.
     * Child-Pugh grade B or C.
  2. Severe renal insufficiency with estimated glomerular filtration rate < 30 ml/min/1.73m2.
  3. Malignant tumor.
  4. A life expectancy of less than 1 year.
* Unsuitable for coronary intervention or long-term antithrombotic therapy

  1. Myocardial bridging located at target lesions.
  2. Major bleeding (BARC type 2 to 5) or active pathological bleeding (including gastrointestinal or genitourinary bleeding) within 3 months,or major surgery within 2 months.
  3. Open surgery is planned within six months after discharge.
  4. Intolerable to double (aspirin plus P2Y12 inhibitor) or single (aspirin or P2Y12 inhibitor) antiplatelet therapy.
  5. History of intracranial hemorrhage.
  6. Pregnant women, lactating women, and women of childbearing potential.
* History of artificial valve replacement.
* History of participating in any other clinical studies or trials within 12 months before the index procedure.
* Participants deemed unsuitable to be enrolled by investigators, such as conditions that may result in protocol nonadherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of a composite of cardiac death, target-vessel myocardial infarction and clinically indicated target vessel revascularization | 12 months
  Incidence of a composite of cardiac death, target-vessel myocardial infarction and clinically indicated target vessel revascularization

SECONDARY OUTCOMES:
Incidence of a composite of peri-procedural complications including cardiac death, perioperative myocardial infarction, acute thrombosis at target vessel and acute occlusion at target vessel | 30 days
  Incidence of a composite of peri-procedural complications including cardiac death, perioperative myocardial infarction, acute thrombosis at target vessel and acute occlusion at target vessel
Incidence of cardiac death | 12 months
  Incidence of cardiac death
Incidence of target-vessel myocardial infarction | 12 months
  Incidence of target-vessel myocardial infarction
Incidence of clinically indicated target vessel revascularization | 12 months
  Incidence of clinically indicated target vessel revascularization
Incidence of a composite of all-cause mortality, nonfatal myocardial infarction, nonfatal stroke, and re-hospitalization | 12 months
  Incidence of a composite of all-cause mortality, nonfatal myocardial infarction, nonfatal stroke, and re-hospitalization
Incidence of major bleeding (Bleeding Academic Research Consortium [BARC] definition, type 2 to 5) | 12 months
  Incidence of major bleeding (Bleeding Academic Research Consortium [BARC] definition, type 2 to 5)
Incidence of net clinical benefit (a composite of cardiac death, target-vessel myocardial infarction, clinically indicated target vessel revascularization and major bleeding) | 12 months
  Incidence of net clinical benefit (a composite of cardiac death, target-vessel myocardial infarction, clinically indicated target vessel revascularization and major bleeding)
Score of Seattle Angina Questionnaire (SAQ) | 1, 6 and 12 months
  SAQ, a 19-item questionnaire that quantifies physical limitations due to angina, any recent change in the severity of angina, the frequency of angina, satisfaction with treatment, and quality of life. SAQ scores range from 0 to 100 and higher scores indicate better health status.
Score of EuroQol Five Dimensions-5L (EQ-5D-5L) | 1, 6 and 12 months
  The EQ-5D-5L questionnaires assesses health in five dimensions (Mobility, Human Autonomy, Current Activities, Pain / Discomfort, Anxiety / Depression), each of which has 5 levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to). Health state index scores generally range from less than 0 to 1, with higher scores indicating higher health utility. The second part of the questionnaire consists of a visual analogue scale on which the patient rates his/her perceived health from 0 to 100.
Quality-adjusted life-years (QALYs) | 12 months
  Quality-adjusted life-years (QALYs)
Total costs | 12 months
  Total costs including the expenditure of hospitalization, physicians, examination, nursing care and medication
Incremental cost-effectiveness ratios (ICER) | 12 months
  The ICER of scheduled DCB compared with conventional DES is defined as the ratio between incremental costs associated with scheduled DCB and the variation in effectiveness. Costs will be measured in Chinese yuan (RMB). Effectiveness will be considered both in terms of life years gained, measured in years, and in terms of quality of life gained, measured in QALY. In the first case, ICER will be measured as RMB/years; in the second, it will be measured as RMB/QALY.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases，Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No